CLINICAL TRIAL: NCT01298466
Title: Open-Labeled European Study To Support The Early Identification Of Patients With Chronic Neuropathic Low Back Pain In Primary Care And To Assess The Effectiveness And Tolerability Of Pregabalin In This Population
Brief Title: Primary Care Identification Of Patients With Chronic Neuropathic Low Back Pain Study
Acronym: PINPOINT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A0081256
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2012-04

CONDITIONS: Low Back Pain; Neuralgia
Keywords: identification; chronic; neuropathic; low back pain; primary care; pregabalin
MeSH Terms: conditions — Low Back Pain; Neuralgia; Bronchiolitis Obliterans Syndrome | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (Experimental): Open label study. All patients fulfilling the protocol inclusion/exclusion criteria will receive pregabalin in a flexible-dosing regimen.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — The investigator will administer pregabalin in a flexible dose-escalation regimen as follows: 150 mg per night for 1 week, 300 mg per day for 1 week, 450 mg per day for 1 week, then 600 mg per day through to the end of the study. Patients may change the dose of medication based on individual response and tolerability as determined by the investigator.

SUMMARY:
A0081256 is a prospective, open-label, multi-centre European study designed to raise awareness and enhance the diagnosis of patients with chronic low back pain with a neuropathic pain component in primary care who are refractory to standard analgesic therapy and/or one treatment for neuropathic pain and evaluate the effectiveness and tolerability of pregabalin in this population. The impact of pregabalin on analgesia, patient satisfaction with treatment, patient anxiety and depression, sleep interference, physical functioning and work productivity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have low back pain with a neuropathic pain component between 3 months and 12 months duration prior to entering the study.
* Patients must have a score of at least 19 on the PainDetect questionnaire and at least 4 on the Standardized Evaluation of Pain (StEP) scale at screening.
* Patients must have a mean pain numerical rating scale (NRS) score of 4 or more during the one week screening period.
* Patients must have failed to respond to standard analgesic therapy (e.g. non-steroidal anti-inflammatory drugs [NSAIDs]) and/or one treatment for neuropathic pain (e.g. tricyclics, serotonin-norepinephrine re-uptake inhibitors [SNRIs]) prior to entering the study).

Exclusion Criteria:

* A diagnosis of depression or a Hospital Anxiety and Depression Scale (HADS) score of > 15 on the depression sub-scale only.
* Patients with a history of renal impairment or who have reduced renal function at baseline (Creatinine Clearance < 60 mL/min).
* Patients who have previously taken pregabalin or gabapentin within 6 months prior to entering the study.
* Patients who have undergone previous surgery for back pain.
* Patients who are using high doses of opioid medication (morphine > 60 mg per day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The change in the daily pain diary (Numerical Rating Scale, NRS) mean pain score at the end of the study (Week 12) compared with baseline. | 12 weeks
The Patients' Global Impression of Change (PGIC) score at the end of the study (Week 12). | 12 weeks

SECONDARY OUTCOMES:
The time to onset of 30% pain reduction (as measured by the NRS mean pain score). | 12 weeks
The change in the Hospital Anxiety and Depression Scale (HADS) score at the end of the study (Week 12) compared with baseline. | 12 weeks
The change in the Sleep Interference Scale score at the end of the study (Week 12) compared with baseline. | 12 weeks
The change in the Lost Work Day Equivalent (LWDE) score at the end of the study (Week 12) compared with baseline. | 12 weeks
The change in the Roland-Morris Disability Questionnaire (RMDQ) score at the end of the study (Week 12) compared with baseline. | 12 weeks
The change in the PainDetect score from baseline versus the change in the Standardized Evaluation of Pain (StEP) score from baseline at the end of the study (Week 12). | 12 weeks
The proportion of patients with a 30% reduction in pain from baseline at study endpoint (as measured by the NRS mean pain score). | 12 weeks
The proportion of patients with a 50% reduction in pain from baseline at study endpoint (as measured by the NRS mean pain score). | 12 weeks
The percentage of primary care physicians who find screening tools useful instruments to support the identification of patients with neuropathic chronic low back pain in daily practice. | 12 weeks
The nature and incidence of adverse events for patients taking 150 mg pregabalin at night as a single dose, either for one week prior to dose escalation or as continued after the option to escalate dose following one week in the study. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081256&StudyName=Primary%20Care%20Identification%20Of%20Patients%20With%20Chronic%20Neuropathic%20Low%20Back%20Pain%20Study